CLINICAL TRIAL: NCT03550417
Title: Evaluation of Medical and Nursing Management for Bronchiectasis
Status: Completed | Type: Observational
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Kathryn Lawton, Principle Investigator, The Queen Elizabeth Hospital
Other Study IDs: QElizabethH
Record Dates: First submitted 2017-04-06; First posted 2018-06-08 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Bronchiectasis
Keywords: disease management; best practice guidelines
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2011 Patients: Evaluation of multidisciplinary management of bronchiectasis compared to the British Thoracic Society Guidelines 2010.
- 2013 Patients: Evaluation of multidisciplinary management of bronchiectasis compared to the British Thoracic Society Guidelines 2010. Comparison of 2011, 2013 cohorts & July16/June17.
- July2016/Jun17 Patients: Evaluation of multidisciplinary management of bronchiectasis compared to the British Thoracic Society Guidelines 2010 & 2014. Comparison of 2011, 2013 cohorts & July16/June17.

SUMMARY:
The purpose of this research is to retrospectively evaluate current clinical care of Bronchiectasis (non-cystic fibrosis [CF]) in adults from a multidisciplinary management perspective. This evaluation aims to address the important gaps in current clinical care in 2011, 2013 and July 2016- Jun2017. The primary outcome of this evaluation is to compare the efficacy of current multidisciplinary clinical practice to the British Thoracic Society (BTS) & Thoracic Society of Australia and New Zealand (TSANZ) guidelines for bronchiectasis. Secondary outcomes of this evaluation will determine the impact of clinical care in 2011, 2013 and July2016-June2017 through quantification of:hospital utilization for using hospital admission data, average length of stay, readmission rates within 28 days, emergency service attendance, outpatient review, exacerbations use of antibiotics, use of Hospital and Home (H@H), number of contacts with the respiratory nursing service and type of contacts with the respiratory nursing service.

DETAILED DESCRIPTION:
Project design: The study will be a 12 month retrospective observational cohort study conducted through a review of medical records, internal respiratory databases and electronic hospital patient record (OACIS, HOMER & EPAS). Participants: Participants in the study will include all patients who have emergency service presentations or admissions to The Queen Elizabeth Hospital (TQEH) with new or existing bronchiectasis in 2011(Jan 1st to Dec 31st). This will be repeated using the same criteria in 2013. An additional year of July2016- Jun2017 has been added for recency of management and to assess if change occurred with introduction of electronic patient record. Data collection: Demographics, clinical data, hospital service utilization, and clinical outcomes such as exacerbation frequency and disease progression. All data will be extracted into a standardized data extraction form, which a random subset will be checked by a second researcher.Analysis of results:Demographic and descriptive data will be given in means + standard deviation and compared using a two-tailed and Student t-test. Categorical variables will be compared using chi-squared or Fisher exact tests, and when appropriate the Mann Whitney U test for non-parametric data. Statistical significance will be determined using an alpha of p <0.05. All analyses will be examined using SPSS software (version x). A subgroup analysis for primary and secondary admission diagnosis will also be performed.

ELIGIBILITY:
Inclusion Criteria: Admission or attendance to emergency services at The Queen Elizabeth hospital with primary or secondary diagnosis of Bronchiectasis in 2011. Repeated using same criteria in 2013 and July2016-June2017

Exclusion Criteria: Patients who do not have bronchiectasis. Patients with traction bronchiectasis. Patients who do not have outpatient follow up. Patients who have follow up by private physicians or other hospitals and records are unavailable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted or attending Emergency Department at The Queen Elizabeth Hospital in 2011, 2013 and July2016-June2017 with primary or secondary diagnosis of bronchiectasis.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with bronchiectasis guideline compliant care | 12 months
  Percentage of patients who meet guideline compliant care for management of bronchiectasis based in TSANZ and BTS guideline recommendations for outpatient management

SECONDARY OUTCOMES:
Number of admissions | 12 months
  Service outcome includes number of emergency department attendance and admissions
Impact of bronchiectasis outpatient management on patient outcomes | 12 months
  Frequency of exacerbation reported in patient case notes (electronic and hard copy) extracted by two respiratory nurses
Number of outpatient (OPD) attendances | 12 months
  Service outcome includes respiratory and all cause OPD attendances
Patient mortality | 0 years up to 4 to 7 years dependent on qualifying year
  Mortality of patients from qualifying admission to present day

CONTACTS AND LOCATIONS:
Overall Officials: Antony Veale, PhD, Study Director — The Queen Elizabeth Hospital

IPD SHARING:
Plan to Share IPD: Yes
Available upon request